CLINICAL TRIAL: NCT00706017
Title: Observational, Safety Study in Subjects Using Levemir® (Insulin Detemir) for the Treatment of Insulin Dependent Type 1 or Type 2 Diabetes Mellitus
Brief Title: Observational Study to Evaluate the Safety of Levemir® in Diabetes
Acronym: PREDICTIVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3518
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Levemir®

SUMMARY:
This observational study is conducted in North America. The aim of this observational study is to evaluate the incidence of adverse events while using Levemir® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes
* Including newly diagnosed not on insulin or insulin analogue treatment
* Selection at the discretion of the physician
* Adult patients with type 1 and 2 diabetes mellitus, and type 1 patients 6 years and older

Exclusion Criteria:

* Current treatment with Levemir®
* Previously enrolled in the study
* Hypersensitivity to Levemir®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from both general and speciality practice settings deemed appropraite to receive Levemir® as new treatment and as part of routine out-patient care by the prescribing physician
Sampling Method: Non-Probability Sample
Enrollment: 2282 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of SADR (serious adverse drug reactions ) incl major hypo (hypoglycaemic events) | during treatment

SECONDARY OUTCOMES:
Glucose control measures | during treatment
Weight | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mexico City, Mexico

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com